CLINICAL TRIAL: NCT03803267
Title: A Comparative Study of Analgesic Effect of Ultrasound Guided Erector Spinae Plane Block Versus Quadratus Lumborum Block for Open Colorectal Cancer Surgeries
Brief Title: Analgesia of Erector Spinae Plane Block Versus Quadratus Lumborum Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MD.18.11.106
Record Dates: First submitted 2019-01-03; First posted 2019-01-14 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Propofol; fentanyl isothiocyanate; Intubation, Intratracheal; Muscle Relaxation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind (participant) study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block (Active Comparator): Patients will receive bilateral ultrasound-guided erector spinae plane block as an adjuvant analgesic technique
  Interventions: Other: Erector spinae plane block; Drug: Propofol; Drug: Fentanyl NCS; Drug: Atracurium Injectable Product; Other: Endotracheal intubation; Drug: Anesthesia Maintenance; Drug: Muscle Relaxation
- Quadratus lumborum block (Active Comparator): Patients will receive bilateral ultrasound-guided quadratus lumborum block as an adjuvant analgesic technique
  Interventions: Other: Quadratus lumborum block; Drug: Propofol; Drug: Fentanyl NCS; Drug: Atracurium Injectable Product; Other: Endotracheal intubation; Drug: Anesthesia Maintenance; Drug: Muscle Relaxation

INTERVENTIONS:
Other: Erector spinae plane block — For each side, the eighth thoracic transverse process will be identified by a linear US transducer (HFL38_10-5 MHz), puncture will be performed in the plane in the craniocaudal direction until the needle contacts the transverse process, and 20 ml of bupivacaine 0.25% and 4 mg dexamethasone will be injected visualizing the hydrodissection. After 30 minutes, the degree of sensory block in the trunk will be assessed by the pinprick test and any undesirable motor weakness will be recorded as a side effect.
  Arms: Erector spinae plane block
Other: Quadratus lumborum block — For each side, shamrock sign with three leaves (psoas major muscle anteriorly, the erector spinae muscle posteriorly and the quadratus lumborum muscle adherent to the apex of the transverse process of the L4 vertebral body) will be identified by a curved array US transducer (6-2MHz), puncture will be performed in-plane, the needle will be advanced through the quadratus lumborum muscle penetrating the ventral proper fascia of the quadratus lumborum muscle, and 20 mL of bupivacaine 0.25% and 4 mg dexamethasone will be injected in that space visualizing the hydrodissection. After 30 minutes, the degree of sensory block in the trunk will be assessed by the pinprick test and any undesired motor weakness will be recorded as a side effect
  Arms: Quadratus lumborum block
Drug: Propofol — Propofol (2 mg/kg)
Drug: Fentanyl NCS — Fentanyl (1µg/Kg)
Drug: Atracurium Injectable Product — atracurium (0.5mg/kg)
Other: Endotracheal intubation — endotracheal intubation
Drug: Anesthesia Maintenance — Inhalational isoflurane in oxygen/air mixture
Drug: Muscle Relaxation — atracurium boluses (0.2 mg/Kg/20 minutes) will be used for maintenance of general anesthesia

SUMMARY:
Colorectal cancer is the third most common cancer worldwide. These patients usually undergo open surgical resection of cancer under general anaesthesia.

The aim of this study is to detect whether the Erector spinae plan block or Quadratus lumborum block will provide the most ideal analgesia for these patients. Erector spinae plan block is a novel analgesic technique that provides both visceral and somatic analgesia due to its communication with the paravertebral space. Quadratus lumborum block is a truncal nerve block usually used for intra-abdominal surgeries. Ultrasound guidance increases the accuracy and safety of both techniques. A local anaesthetic mixture of Bupivacaine 0.25% and dexamethasone will be used for both techniques.

DETAILED DESCRIPTION:
Erector spinae plane block and quadratus lumborum block are analgesic techniques suitable for open colorectal cancer surgeries. postoperative pain score, serum levels of biomarkers of stress (cortisol and CRP), primary hemodynamics, time to first rescue analgesic request, the total amount of rescue analgesic consumption and postoperative nausea and vomiting are the parameters of comparison between both techniques.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I or II
* Body mass index from 18.5 to 35 Kg/m2

Exclusion Criteria:

* Body mass index more than 35 Kg/m2.
* Severe or uncompensated cardiovascular disease.
* Severe renal disease.
* Severe hepatic disease.
* Severe endocrinal disease.
* Pregnancy.
* Postpartum.
* Lactating females
* Allergy to one of the agents used.
* Refusal to participate in the study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score | From 1 day before the surgery to the 2 days after surgery
  The intensity of pain indicated by a segmented numeric scale in which a respondent selects a whole number (0-100 integers) that best reflects his/her pain as 0-30 for mild pain, 30-60 for moderate pain and 60-100 for sever pain

SECONDARY OUTCOMES:
Systolic Blood Pressure | One hour before induction of general anesthesia, every 10 minutes till end of surgery, every 4 hours till end of the first 24 hours postoperatively, then every 8 hours till end of the next 24 hours
  The pressure in the arteries during contraction of the heart
Mean Blood Pressure | One hour before induction of general anesthesia, every 10 minutes till end of surgery, every 4 hours till end of the first 24 hours postoperatively, then every 8 hours till end of the next 24 hours
  : The average pressure in the arteries during one cardiac cycle. It is a better indicator for vital organs' perfusion than the systolic pressure
Heart rate | One hour before induction of general anesthesia, every 10 minutes till end of surgery, every 4 hours till end of the first 24 hours postoperatively, then every 8 hours till end of the next 24 hours
  The number of heart beats per minute. A lower heart rate at rest implies a more efficient heart function, better cardiovascular fitness and less stress
Time to first rescue analgesic request | Up to 48 postoperative hours
  The time elapsed from termination of performing each block till the patient's request for analgesia. It resembles the duration of analgesia
Peripheral oxygen saturation | One hour before induction of general anesthesia, every 10 minutes till end of surgery, every 4 hours till end of the first 24 hours postoperatively, then every 8 hours till end of the next 24 hours
  An estimate of oxygenated hemoglobin concentration in blood. It is measured by pulse oximeter device
Total amount of rescue analgesic consumption | From the time of first analgesic request till the end of the first 24 hours, then till the end of the next 24 hours postoperatively
  The total amount of morphine consumed by the patient for pain relief over the 48 hours postoperatively
Postoperative nausea and vomiting intensity score | Immediately after recovery, every 4 hours till end of the first 24 hours postoperatively, then every 8 hours till end of the next 24 hours
  Postoperative Nausea and Vomiting Intensity Scale: A scale that evaluates postoperative nausea and vomiting. It equals severity of nausea (1=mild, 2= moderate, 3= sever) x pattern of nausea (1=varying, 2= constant) x duration of nausea (in hours). At any time, if it is < 50 or vomiting occurs once or twice, it is clinically unimportant (good outcome). If it is ≥50 or vomiting occurs 3 or more times, it is clinically important (bad outcome). The sum of all values will quantify the entire period of the study.
Cortisol | At 9 Am, 1 hour after induction of general anesthesia, 1st, 24th and 48th hours postoperatively
  A steroid hormone secreted by adrenal cortex in response to stress and hypoglycemia
Serum C-reactive protein (CRP) | On hospital admission, 1 hour after induction of general anesthesia, 1st, 24th and 48th hours postoperatively
  A protein synthetized by hepatocytes in response to systemic inflammation or tissue damage

CONTACTS AND LOCATIONS:
Overall Officials: Amer A Attieh, MD, Study Chair — Professor; Mohammed A Ghanem, MD, Study Director — Associate Professor
Locations (1):
- Amer A Attieh, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided